CLINICAL TRIAL: NCT02327325
Title: Physical Activity for Older Adults With Chronic Low Back Pain: PACe-LBP
Brief Title: Physical Activity for Older Adults Chronic Low Back Pain
Acronym: PACe-LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E1569-P
Record Dates: First submitted 2014-12-08; First posted 2014-12-30 (Estimated); Results first posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Exercise; Cognitive Behavioral Therapy; Aged
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Exercise; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Physical Activity Only (Experimental): 12-week home-based physical activity program with telephone support. Delivered by a physical therapist and exercise counselor. Comprehensive program including stretching, strengthening and aerobic activity.
  Interventions: Behavioral: Physical Activity
- Physical Activity + Cognitive Behavioral Therapy (Experimental): 12-week combined home-based physical activity and cognitive behavioral program with telephone support. Delivered by a physical therapist and exercise counselor. Comprehensive physical activity program including stretching, strengthening and aerobic activity. Cognitive behavioral component includes training in multiple skills for managing pain.
  Interventions: Behavioral: Physical Activity; Behavioral: Cognitive Behavioral Therapy
- Wait List Control Group (No Intervention): Will receive the physical activity only or physical activity + cognitive behavioral therapy (based on participant choice) after completing all follow-up assessments.

INTERVENTIONS:
Behavioral: Physical Activity — 12-week home-based physical activity program with telephone support. Delivered by a physical therapist and exercise counselor. Comprehensive program including stretching, strengthening and aerobic activity.
  Arms: Physical Activity + Cognitive Behavioral Therapy; Physical Activity Only
Behavioral: Cognitive Behavioral Therapy — Telephone-based training in multiple skills for managing low back pain.
  Arms: Physical Activity + Cognitive Behavioral Therapy

SUMMARY:
Chronic low back pain (cLBP) is one of the most common and disabling conditions among US military Veterans. Although physical activity can improve cLBP outcomes, the majority of Veterans with cLBP are inactive. Therefore the VA is in need of effective programs that can help older Veterans with cLBP to increase their physical activity and improve associated outcomes. This is particularly relevant for older Veterans with cLBP who are at greater risk for functional limitations. The proposed project will be a pilot study of a telephone-based physical activity program or physical activity combined with cognitive behavioral pain management for older adult Veterans with cLBP. Older Veterans are of particular interest because prior studies of physical activity for cLBP have not addressed this vulnerable patient group. This study will also inform the VA about whether certain patients with cLBP, who have greater pain sensitivity, may benefit from other treatment to supplement a physical activity program.

DETAILED DESCRIPTION:
Chronic low back pain (cLBP) is one of the most common and disabling conditions among US military Veterans, and the prevalence is rising even more rapidly than other chronic conditions such as diabetes and hypertension. Studies have shown that physical activity (PA) can improve outcomes in patients with cLBP, but a major gap in this research is the lack of studies focusing on older adults; patient samples have been primarily middle-aged and have included few patients' age 65 years. Therefore, the investigators' lack an evidence base for the feasibility and effectiveness of PA interventions in this vulnerable group of patients with cLBP. This is particularly important given the accumulating evidence showing that older adults with cLBP have significant lower extremity functional limitations, resulting in difficulty performing necessary daily tasks. Another area of limited investigation among older adults with cLBP is whether there is added benefit of incorporating cognitive behavioral therapy for pain management (CBT-P) skills with PA interventions. CBT-P can help to restructure pain perception and improve pacing of PA. Some patients with cLBP do not respond favorably to isolated PA interventions, and it is possible that heightened pain sensitization may underlie this lack of response in some patients. Since CBT-P has been shown to alter pain processing, older adults with cLBP who have greater pain sensitization may respond better to a program that combines PA and CBT-P (vs. PA alone); however, this has not been studied. This information has practical implications for a larger trial to determining whether a subset of patients with greater central pain sensitivity may need additional intervention to supplement a PA program.

The investigators will conduct a pilot study of a 12-week home-based PA and PA + CBT-P programs, both with weekly telephone support, compared with a waiting list control group. Participants will be 60 older Veterans (age 65) with cLBP. Enrollment of participants will occur via referrals from geriatric and primary care clinics at the Durham VAMC. The PA program will be comprehensive, including stretching, strengthening, and aerobic activities, and the specific types and intensities of the activities will be geared toward older adults. The CBT-P program will include five different skills, woven into the telephone-based sessions, with specific application to PA and cLBP. Both interventions will be jointly delivered by a physical therapist and exercise counselor, who has complementary areas of expertise (e.g., training in clinical exercise prescription and motivational interviewing skills to encourage PA adherence, respectively). Telephone calls will involve patient-specific goal-setting and address barriers to PA and CBT-P skills. Participants will receive a booklet with instructions and photographs for stretching and strengthening exercises, as well as an exercise video appropriate for older adults with cLBP. Participants in the combined intervention will also receive written and audio instructions regarding CBT-P skills. Feasibility measures will include the proportion of completed intervention calls, adherence to home-based PA recommendations and CBT-P skills use, and participant feedback on the programs. Outcomes will be assessed at baseline and 12-week follow-up. Primary measures of efficacy will be assessments of general physical function, both objective and self-reported (PROMIS Health Assessment Questionnaire). Secondary outcomes will include measures cLBP-specific pain and disability. Central pain sensitivity will be assessed via Pain Pressure Threshold (PPT) testing and the Central Sensitization Inventory (CSI). Statistical analyses will include comparison of baseline and follow-up outcomes across study groups, as well as examination of potential trends for differential intervention response according to baseline PPT and CSI scores.

ELIGIBILITY:
Inclusion Criteria:

1. Self-report having had lower back pain on most days for greater than three months.
2. Can complete a 10 second semi-tandem stand and walk 8' in 6.0 seconds.
3. Report they are not satisfied with their current state of functional ability, based on reporting "dissatisfied" with at least one aspect of physical function on the Satisfaction with Physical Function Scale.
4. Can safely participate in the intervention based upon the physical therapist baseline examination and clinical expertise.

Exclusion Criteria:

1. unilateral or bilateral sciatica that physical therapist determines could make the study intervention unsafe or inappropriate; isolated coccyx pain (based on self-report at screener);
2. dementia or other significant cognitive impairment;
3. movement or motor neuron disorders (e.g., Parkinson's Disease, Multiple Sclerosis, Amyotrophic Lateral Sclerosis);
4. rheumatoid arthritis, fibromyalgia, or other systemic rheumatic disease;
5. hospitalization for a stroke, myocardial infarction, heart failure, or coronary artery revascularization in the past 3 months;
6. significant hearing impairment (must be able to talk on the telephone);
7. psychosis or current, uncontrolled substance abuse disorder;
8. any other health conditions determined by the study team to be contraindications to performing mild to moderate home exercises.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Dominick Allen, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goode AP, Taylor SS, Hastings SN, Stanwyck C, Coffman CJ, Allen KD. Effects of a Home-Based Telephone-Supported Physical Activity Program for Older Adult Veterans With Chronic Low Back Pain. Phys Ther. 2018 May 1;98(5):369-380. doi: 10.1093/ptj/pzy026. PMID 29669086

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Physical Activity Only | Physical Activity + Cognitive Behavioral Therapy | Wait List Control Group
Started | 20 | 20 | 20
Completed | 19 | 16 | 15
Not Completed | 1 | 4 | 5
Not completed — Withdrawal by Subject | 1 | 4 | 4
Not completed — Excluded by Study Team | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Activity Only | Physical Activity + Cognitive Behavioral Therapy | Wait List Control Group | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (3.5) | 69.5 (4.0) | 71.9 (6.5) | 70.3 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 19 | 18 | 19 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 19 | 20 | 20 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 11 | 9 | 31
  White | 8 | 9 | 11 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Education Level [Count of Participants; unit: Participants]
  At least some college | 13 | 10 | 8 | 31
  High school or technical school | 7 | 10 | 12 | 29
Employment Status [Count of Participants; unit: Participants]
  Disabled | 7 | 8 | 6 | 21
  Other | 13 | 12 | 14 | 39
Marital Status [Count of Participants; unit: Participants]
  Married | 9 | 13 | 16 | 38
  Other | 11 | 7 | 4 | 22
Household Financial Status [Count of Participants; unit: Participants] — Low income defined as self-report of "just meeting basic expenses" or "don't have enough to meet basic expenses". Population: Two participants declined to answer.
  Participants
    number analyzed (Participants) | 20 | 19 | 19 | 58
    Low income | 4 | 6 | 6 | 16
    Other | 16 | 13 | 13 | 42

OUTCOME MEASURES:

1. Primary Outcome: Timed Get-Up-And Go
Description: This test requires the participants to stand from a standard arm chair, walk 3 meters and then return to sitting in the same chair. Greater number of seconds is associated with poorer physical function. Therefore, a positive change from baseline to follow-up means worsening function; a negative change (e.g., lower score at follow-up than at baseline) indicated improving function.
Time Frame: Change from baseline to 12-week follow-up
Population: The analysis populations includes all participants except for one who was unable to stand without assistance and declined to perform this test at both baseline and follow-up.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Physical Activity Only | Physical Activity + Cognitive Behavioral Therapy | Wait List Control Group
Number analyzed (Participants) | 20 | 19 | 20
seconds | -1.84 [-4.01 to 0.33] | -2.15 [-4.52 to 0.21] | 1.11 [-1.24 to 3.47]
Statistical Analysis 1: Comparison: Physical Activity Only vs Wait List Control Group; This is the comparison between physical activity only and the wait list group. Rejection of the null hypothesis means that the physical activity group had greater improvement than the wait list group; Test type: Superiority; p = 0.08, Mixed Models Analysis; Mean Difference (Final Values) = -2.94, 95% CI 2-sided [-6.24 to 0.35]
Statistical Analysis 2: Comparison: Physical Activity + Cognitive Behavioral Therapy vs Wait List Control Group; This is the comparison of the PA & CBT group to the wait list group. Rejection of the null hypothesis means that the PA + CBT group was superior on this outcome to the wait list group; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = -3.26, 95% CI 2-sided [-6.69 to 0.06]

2. Primary Outcome: PROMIS Health Assessment Questionnaire
Description: Self-reported physical function/disability measure that captures both activities of daily living and instrumental activities of daily living. It consists of 20-items scored on a 0-3 scale with a summed 0-100-unit scale. Higher scores are associated with worse function. Therefore a positive change score indicates worsening over time; negative change score (e.g., lower score at follow-up) indicates improvement.
Time Frame: Change from baseline to 12-week follow-up
Population: 18 participants are missing data from this questionnaire because they entered a response of "don't know" for one or more items, and there were not adequate instructions for scoring the questionnaire with the missing data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Physical Activity Only | Physical Activity + Cognitive Behavioral Therapy | Wait List Control Group
Number analyzed (Participants) | 16 | 11 | 15
units on a scale | -2.90 [-7.22 to 1.43] | -0.89 [-6.36 to 4.57] | 3.21 [-1.61 to 8.02]
Statistical Analysis 1: Comparison: Physical Activity Only vs Wait List Control Group; This is the comparison of the PA only group with the wait list control. Rejection of the null hypothesis means that the PA group was superior to the wait list group; Test type: Superiority; p = 0.07, Mixed Models Analysis; Mean Difference (Net) = -6.11, 95% CI 2-sided [-12.85 to 0.64]
Statistical Analysis 2: Comparison: Physical Activity + Cognitive Behavioral Therapy vs Wait List Control Group; This is the comparison of the PA + CBT only group with the wait list control. Rejection of the null hypothesis means that the PA + CBT group was superior to the wait list group; Test type: Superiority; p = 0.28, Mixed Models Analysis; Mean Difference (Final Values) = -4.10, 95% CI 2-sided [-11.69 to 3.48]

3. Secondary Outcome: Patient Specific Functional Scale
Description: This measure captures items that are specific functional tasks that may be missed on standardized questionnaires. The measure consists of 3 items specifically provided by the patient. Each item provided by the patient is score from a 0 (Unable to perform task) to 10 (able to complete the activity without difficulty) scale. Higher change scores from baseline to follow up indicate more improvement (total range 0-30).
Time Frame: Change from baseline to 12-week follow-up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Physical Activity Only | Physical Activity + Cognitive Behavioral Therapy | Wait List Control Group
Number analyzed (Participants) | 20 | 20 | 20
units on a scale | 3.72 [0.89 to 6.55] | 3.00 [-0.04 to 6.04] | 0.08 [-3.12 to 3.39]
Statistical Analysis 1: Comparison: Physical Activity Only vs Wait List Control Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.097, Mixed Models Analysis; Mean Difference (Final Values) = 3.64, 95% CI 2-sided [-0.69 to 7.96]
Statistical Analysis 2: Comparison: Physical Activity + Cognitive Behavioral Therapy vs Wait List Control Group; This is the comparison of the PA+CBT group with the wait list control. Rejection of the null hypothesis means that the PA+CBT group was superior to the wait list group; Test type: Superiority; p = 0.196, Mixed Models Analysis; Mean Difference (Final Values) = 2.91, 95% CI 2-sided [-1.55 to 7.39]

4. Secondary Outcome: Roland-Morris Disease Specific Disability Questionnaire
Description: 24-item self-report measure of low back pain-specific disability. Higher scores indicate worse function, with a range of 0=no disability to 24=maximum disability measured by the scale. Therefore a positive change score indicates worsening. A negative change score (e.g., lower score at follow-up) indicates improvement.
Time Frame: Change from baseline to 12-week follow-up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Physical Activity Only | Physical Activity + Cognitive Behavioral Therapy | Wait List Control Group
Number analyzed (Participants) | 20 | 20 | 20
units on a scale | -3.21 [-5.01 to -1.41] | -1.11 [-3.05 to 0.83] | 0.89 [-1.11 to 2.88]
Statistical Analysis 1: Comparison: Physical Activity Only vs Wait List Control Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.01, Mixed Models Analysis; Mean Difference (Final Values) = -4.10, 95% CI 2-sided [-6.85 to -1.34]
Statistical Analysis 2: Comparison: Physical Activity + Cognitive Behavioral Therapy vs Wait List Control Group; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.17, Mixed Models Analysis; Mean Difference (Final Values) = -1.99, 95% CI 2-sided [-4.85 to 0.86]

5. Secondary Outcome: Satisfaction With Physical Function Scale
Description: This is a validated 5-item questionnaire that assesses patients' satisfaction with their ability to complete basic functional tasks that are often affected by lower extremity OA, including stair-climbing, walking, doing housework (light and heavy, and lifting and carrying. All items are rated on a 7-point scale ranging from Very Dissatisfied (-3) Very Satisfied (+3). A positive change score indicates improvement, and a negative change score indicates worsening.
Time Frame: Change from baseline to 12-week follow-up
Population: 6 participants are missing data from this questionnaire because they entered a response of "don't know" for one or more items, and there were not adequate instructions for scoring the questionnaire with the missing data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Physical Activity Only | Physical Activity + Cognitive Behavioral Therapy | Wait List Control Group
Number analyzed (Participants) | 18 | 18 | 18
units on a scale | 3.11 [-0.23 to 6.46] | 3.06 [-0.68 to 6.81] | 2.96 [-0.58 to 6.49]
Statistical Analysis 1: Comparison: Physical Activity Only vs Wait List Control Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.95, Mixed Models Analysis; Median Difference (Final Values) = 0.16, 95% CI 2-sided [-4.86 to 5.19]
Statistical Analysis 2: Comparison: Physical Activity + Cognitive Behavioral Therapy vs Wait List Control Group; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.97, Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-7.07 to 1.07]

ADVERSE EVENTS:
Arm/Group | Physical Activity Only | Physical Activity + Cognitive Behavioral Therapy | Wait List Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activity Only (N=20) | Physical Activity + Cognitive Behavioral Therapy (N=20) | Wait List Control Group (N=20)
Hospitalization (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Hospitalization due to fall resulting in multiple fractures
Hospitalizatoin (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Hospitalization for acute renal failure injury secondary to volume depletion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT02327325/Prot_SAP_000.pdf